CLINICAL TRIAL: NCT07242560
Title: Factors Associated With Infection Development in Epidural Catheter and Port Applications in a University Pain Clinic: A Retrospective Cohort Study
Brief Title: Epidural Catheter and Port-Related Infections in Pain Clinic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Mesut Bakır (Other)
Responsible Party: Sponsor-Investigator, Mesut Bakır, Assoc. Prof. Dr. Mesut Bakır, Mersin University Faculty of Medicine, Department of Algology, Mersin University
Organization: Mersin University (Other)
Other Study IDs: Mersin-ALG-ECPI-2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Epidural Catheter-Related Infection; Hospital-Acquired Infection; Procedural Complication
Keywords: Epidural catheter; Epidural port; Infection; Pain clinic; Interventional pain management
MeSH Terms: conditions — Cross Infection; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural Catheter Group: Patients who underwent epidural catheter insertion for pain management between January 2002 and December 2022 at the Mersin University Pain Clinic. Data include catheter duration, insertion site, indication, and culture results.
- Epidural Port Group: Patients who received epidural port placement for long-term analgesic management during the same period. Data include port type, indication, duration of use, and infection outcomes.

SUMMARY:
This retrospective observational study aims to evaluate the incidence and risk factors of infection associated with epidural catheter and port applications performed in the Pain Clinic of Mersin University Faculty of Medicine. Data from patients who underwent epidural catheter or port placement between January 2002 and January 2025 will be analyzed.

Demographic data, catheter duration, insertion level, type of device, clinical indication, and microbiological culture results will be examined to determine factors influencing infection development. The study seeks to identify common pathogens and assess potential relationships between procedural characteristics and infection risk.

The ultimate goal of this research is to contribute to improving infection prevention strategies and ensuring patient safety in interventional pain management practices.

DETAILED DESCRIPTION:
This retrospective cohort study investigates the factors associated with infection development following epidural catheter and port applications performed in the Pain Clinic of Mersin University Faculty of Medicine between January 2002 and January 2022. Data collection has been completed, and the final data analysis is expected to be finalized by November 30, 2025.

Epidural catheterization and port placement are frequently performed interventional pain management procedures used for postoperative and chronic cancer pain treatment. Despite their clinical utility, these procedures carry a risk of infection that can lead to serious complications, including epidural abscess, meningitis, or systemic sepsis.

The study retrospectively reviews 351 cases from institutional archives. Demographic data (age, sex, diagnosis), procedural details (catheter duration, insertion level, anatomical site, indication, brand), and infection outcomes (presence of infection, culture results, and isolated microorganisms) are analyzed.

Primary outcome is the incidence of infection associated with epidural catheter or port use. Secondary outcomes include identifying risk factors such as catheter duration, insertion site, clinical indication, and the distribution of isolated pathogens. Statistical analyses are conducted using appropriate parametric or non-parametric tests, and p < 0.05 is considered significant.

The findings of this study are expected to contribute to improving infection prevention strategies and clinical protocols for safer interventional pain management practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Patients who underwent epidural catheter or epidural port application at Mersin University Pain Clinic between January 1, 2002 and January 1, 2025.
* Complete clinical records including demographic data, procedural details, and culture results available for review.

Exclusion Criteria:

* Patients with incomplete or missing procedural or infection data.

Patients whose records do not include culture or infection status documentation.

Patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Pain Clinic of Mersin University Faculty of Medicine who received epidural catheter or port applications for pain management between 2002 and 2025.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Infection Associated With Epidural Catheter or Port Use | From date of catheter or port placement until device removal or completion of follow-up (within study period January 2002-January 2025).
  The proportion of patients who developed infection following epidural catheter or port placement, confirmed either clinically or microbiologically (positive culture from catheter tip or port site).

SECONDARY OUTCOMES:
Risk Factors Associated With Infection Development | Throughout the duration of catheter or port use, within the study period (January 2002-January 2025).
  Evaluation of demographic and procedural variables (e.g., catheter duration, insertion site, indication, comorbidities) and their association with infection occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Bakır, Assoc. Prof, Principal Investigator — Mersin University Faculty of Medicine, Pain Clinic
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective study based on de-identified patient records. No individual participant data (IPD) will be shared. Only aggregated results may be published in scientific journals.

REFERENCES:
- [Background] Horlocker TT, Wedel DJ. Infectious complications of regional anesthesia. Best Pract Res Clin Anaesthesiol. 2008 Sep;22(3):451-75. doi: 10.1016/j.bpa.2008.06.003. PMID 18831298
- [Background] Domingues C, Goncalves L, Laranjo M, Santos T, Goncalves D, Goncalves L, Barros AC, Marrao G, Castro R, Valente E. Epidural Catheter Bacterial Colonization and Infection in a Secondary Portuguese Hospital Setting. Cureus. 2024 Oct 26;16(10):e72428. doi: 10.7759/cureus.72428. eCollection 2024 Oct. PMID 39588402